CLINICAL TRIAL: NCT02759991
Title: An Effectiveness Trial (Phase IV) to Evaluate Protection of Pregnant Women by Hepatitis E Virus (HEV) Vaccine in Bangladesh and Risk Factors for Severe HEV Infection.
Brief Title: Effectiveness Trial to Evaluate Protection of Pregnant Women by Hepatitis E Vaccine in Bangladesh.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Norwegian Institute of Public Health (Other Government)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); Sykehuset Innlandet HF (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 61067
Record Dates: First submitted 2016-03-21; First posted 2016-05-03 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2020-10

CONDITIONS: Hepatitis E Infection
Keywords: Hepatitis E virus; Viral Hepatitis Vaccines
MeSH Terms: interventions — hecolin; Hepatitis B Vaccines; Vaccines

STUDY DESIGN:
Intervention Model Description: 1. Pilot study completed in 2017 with 100 participants, 50 women and 50 men aged 16-39, randomized to be vaccinated with either 2 doses of Hecolin or Hepa-B. These 100 participants are not included in the main trial.
  2. Main clinical trial designed to enroll 20.745 women aged 16-39 years living in Matlab area. All participants randomized to be vaccinated with either Hecolin or Hepa-B three doses.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HEV vaccine (Active Comparator): Hecolin, 0.6 ml intramuscular injection day 0, 1 month and 6 months.
  Interventions: Drug: Hecolin
- HBV vaccine (Placebo Comparator): Hepa-B, 1 ml intramuscular injection day 0, 1 month and 6 months.
  Interventions: Drug: Hepa-B

INTERVENTIONS:
Drug: Hecolin — 0.6ml Hecolin vaccine im. on day 0, 1 month and 6 months.
  Other Names: HEV 239
  Arms: HEV vaccine
Drug: Hepa-B — 1ml Hepa-B vaccine im. on day 0, 1 month and 6 months.
  Other Names: Hepatitis B virus (HBV) vaccine
  Arms: HBV vaccine

SUMMARY:
The aim of the study is to determine the effectiveness of hepatitis E virus vaccine given in women of child bearing age in preventing HEV disease during pregnancy among women in rural Bangladesh.

DETAILED DESCRIPTION:
Hepatitis E virus (HEV) infection is endemic in Bangladesh, causing severe or fatal complications in pregnant women. This GLOBVAC funded project aims to assess the safety, feasibility, acceptability, immunogenicity, effectiveness, and cost-effectiveness of the HEV vaccine (Hecolin, Innovax, China) when given women of childbearing age in a rural area in Bangladesh (Matlab). The vaccine has been shown to be both effective and safe in the general adult population in China, but there is insufficient data about its efficacy among pregnant women, the group with most to gain from vaccination.

The research plan has been carefully designed and will be conducted by a multidisciplinary team of researchers at International Centre for Diarrhoeal Disease Research (iccdr,b) in Bangladesh and the Norwegian Institute of Public Health and Innlandet Hospital Trust in Norway. Over a period of 2 years, 20,745 non-pregnant women will be recruited and will receive either the hepatitis E vaccine or a hepatitis B vaccine (control group). All women who develop hepatitis E symptoms will be tested for the disease. Those who become pregnant during the study will also be checked and tested during regular home visits. Clinical outcomes and vaccine adverse events will be closely monitored.

In order to evaluate the initial safety profile and immunogenicity of the vaccine, a pilot study was completed during summer 2017. A total of 100 non-pregnant females and males, aged 16-39, were enrolled and randomly received either the hepatitis E vaccine or a hepatitis B vaccine. Participants were vaccinated on day 0 and day 30, and blood, dried blood spots (DBS) and saliva samples were collected on day 0 and day 60 for use in laboratory assay validation and serological and cellular immunogenicity analyses. Following each vaccination, home visits were carried out for 7 days to record adverse reactions. No serious adverse reactions were observed, and only a few mild local adverse reactions were recorded which all resolved without sequela. Preliminary immunogenicity results, showed that 44 participants had seroconverted (HEV), after just two doses of the vaccine. Furthermore, during this pilot study the implementation of protocols and procedures for all stages of the trial were tested in preparation for the start of the main trial.

Additionally, hepatitis surveillance in Matlab has been initiated in order to establish an HEV surveillance system. All women aged 16-39 are included in the surveillance, and requested to contact icddr,b staff if they experience jaundice of any duration, or other symptoms of hepatitis. Patients admitted to Matlab hospital have a blood sample taken for hepatitis diagnostics, and acute HEV cases are investigated virologically, clinically and immunologically. Household visits occur bi-weekly to document any possible hepatitis cases.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 16-39 years
* Living in Matlab area

Exclusion Criteria:

* Pregnancy
* Allergic to vaccine components
* Serious chronic diseases
* Acute illness

Ages: 16 Years to 39 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 19460 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Effectiveness of HEV vaccine in preventing HEV diseases among women in Bangladesh | 2 years
  To determine the effectiveness of hepatitis E virus (HEV) vaccine in preventing HEV disease during pregnancy among women in rural Bangladesh

SECONDARY OUTCOMES:
To determine the safety of HEV vaccine in Bangladeshi women of childbearing age | 2 years
  Number of participants with adverse events related to vaccination as assessed by CTCAE v4.0
To determine the immunogenicity of HEV vaccine in Bangladeshi women of childbearing age | 2 years
  Number of participants who seroconvert after three doses
Effectiveness of HEV vaccine in preventing HEV disease in non-pregnant Bangladeshi women of childbearing age | 2 years
  To determine the effectiveness of hepatitis E virus (HEV) vaccine in preventing HEV disease in participants
Estimate serological correlates of protection | 2 years
  Assess the anti-HEV IgG levels before and one month after the last dose of vaccine for primary vaccine response and record if any HEV disease occurs.
Assess the feasibility, acceptability and cost-effectiveness of HEV vaccination of women of childbearing age in rural Bangladesh | 2 years
  Analyse cost per disability, adjusted life year and quality adjusted life year
Investigate acute HEV cases virologically, clinically and immunologically in relation to outcome. | 2 years
  Examine acute HEV cases in relation to severity of illness and immunological responses

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Dudman, MD, PhD, Principal Investigator — Norwegian Institute of Public Health; K Zaman, PhD, Principal Investigator — International Centre for Diarrhoeal Disease Research, Bangladesh, Centre for Child and Adolescent Health
Locations (1):
- International Centre for Diarrhoeal Disease Research, Bangladesh, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Overbo J, Dembinski JL, Nilsen TR, Sriranganathan V, Dimova-Svetoslavova VP, Aziz A, Zaman K, Julin CH, Qadri F, Stene-Johansen K, Bhuiyan TR, Haque W, Dudman S. Cellular and Humoral Immune Profiles After Hepatitis E Vaccination and Infection. Viruses. 2025 Jun 26;17(7):901. doi: 10.3390/v17070901. PMID 40733519
- [Derived] Aziz AB, Dudman S, Julin CH, Ahmmed F, Stene-Johansen K, Sandbu S, Overbo J, Dembinski JL, Wisloff T, Rana S, Basunia AH, Haque W, Qadri F, Zaman K, Clemens JD. Receipt of hepatitis E vaccine and fetal loss in rural Bangladesh: further analysis of a double-blind, cluster-randomised, controlled trial. Lancet Glob Health. 2024 Aug;12(8):e1300-e1311. doi: 10.1016/S2214-109X(24)00193-1. PMID 39030061
- [Derived] Zaman K, Julin CH, Aziz AB, Stene-Johansen K, Yunus M, Qadri F, Gurley ES, Sandbu S, Overbo J, Dembinski JL, Laake I, Bhuiyan TR, Rahman M, Haque W, Khanam M, Clemens JD, Dudman S. Safety and effectiveness of a recombinant hepatitis E vaccine in women of childbearing age in rural Bangladesh: a phase 4, double-blind, cluster-randomised, controlled trial. Lancet Glob Health. 2024 Aug;12(8):e1288-e1299. doi: 10.1016/S2214-109X(24)00192-X. PMID 39030060
- [Derived] Overbo J, Aziz A, Zaman K, Clemens J, Halle Julin C, Qadri F, Stene-Johansen K, Biswas R, Islam S, Rahman Bhuiyan T, Haque W, Sandbu S, Elahee ME, Ali M, Dembinski JL, Dudman S. Immunogenicity and safety of a two-dose regimen with hepatitis E virus vaccine in healthy adults in rural Bangladesh: A randomized, double-blind, controlled, phase 2/pilot trial. Vaccine. 2023 Jan 27;41(5):1059-1066. doi: 10.1016/j.vaccine.2022.12.064. Epub 2023 Jan 2. PMID 36599736
- [Derived] Zaman K, Dudman S, Stene-Johansen K, Qadri F, Yunus M, Sandbu S, Gurley ES, Overbo J, Julin CH, Dembinski JL, Nahar Q, Rahman A, Bhuiyan TR, Rahman M, Haque W, Khan J, Aziz A, Khanam M, Streatfield PK, Clemens JD. HEV study protocol : design of a cluster-randomised, blinded trial to assess the safety, immunogenicity and effectiveness of the hepatitis E vaccine HEV 239 (Hecolin) in women of childbearing age in rural Bangladesh. BMJ Open. 2020 Jan 19;10(1):e033702. doi: 10.1136/bmjopen-2019-033702. PMID 31959609

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/91/NCT02759991/Prot_SAP_ICF_000.pdf